CLINICAL TRIAL: NCT07091149
Title: Digital Cognitive Behavioral Treatment of Insomnia in Youth: An RCT Examining Feasibility, Acceptability, and Efficacy of NiteCAPP Jr
Acronym: NiteCAPP JR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY006258
Record Dates: First submitted 2025-04-10; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: dCBTi; digital intervention; insomnia; children
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either CBT-I or a waitlist control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I (Experimental): Immediate CBT-I for typically developing children using a 4-session digital intervention.
  Interventions: Behavioral: CBT-I
- Waitlist Control (Other): Participants in the waitlist control will have delayed treatment (4 weeks later).
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — Cognitive behavioral therapy for insomnia

SUMMARY:
The proposed pilot will examine feasibility, acceptability, and preliminary efficacy of a digital CBT-I tailored for school-aged children.

DETAILED DESCRIPTION:
This is a pilot study to examine feasibility, acceptability, and preliminary efficacy of a digital CBT-I tailored for school-aged children aged 6-12 with insomnia and their caregiver(s) compared to a waitlist control.

ELIGIBILITY:
Inclusion Criteria:

Child inclusion:

1. 6-12 yrs
2. Verbal IQ > 70 (to ensure verbal skills are sufficient to participate in treatment)
3. participation of child's parent or legal guardian living in the same home
4. child diagnosed with insomnia, 5) willing to accept random assignment.

Insomnia:

1) insomnia complaints for 3+ months by child report or caregiver observation that consist of (a) difficulties falling asleep, staying asleep, and/or waking up too early, (b) daytime dysfunction (mood, cognitive, social, occupational) due to insomnia, and (c) Pediatric Insomnia Severity Index score >8

Caregiver inclusion:

1. ability to read and understand English at the 5th grade level
2. willing to accept random assignment.

Exclusion Criteria:

Child exclusion:

1. child unable to provide informed consent or child unable to provide assent
2. child unwilling to accept random assignment
3. child participation in another randomized research project
4. child unable to complete forms or implement treatment procedures due to cognitive impairment
5. child untreated medical comorbidity including other sleep disorders (e.g., apnea, epilepsy, psychotic disorders, suicidal ideation/intent, [frequent] parasomnias)
6. child psychotropic or other medications that alter sleep with the exceptions of stimulants, sleep medications, and/or melatonin as described in #7 (see Notes below for details)
7. child stimulants, sleep medications (prescribed or OTC), and/or melatonin within the last 1 month (unless stabilized on medication for 3+ months)
8. child participation in non-pharmacological treatment (including CBT) for sleep outside current trial
9. child other conditions adversely affecting trial participation.

Caregiver exclusion criteria:

1. unable to provide informed consent
2. unwilling to accept random assignment
3. caregiver participation in another randomized research project
4. unable to complete forms or implement treatment procedures due to cognitive impairment
5. caregiver participation in non-pharmacological treatment (including CBT) for sleep outside current trial

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Electronic Sleep Diaries - Child | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Primary: child sleep onset latency (lights-out until sleep onset) and total sleep time. All other sleep diary variables are secondary (e.g., sleep efficiency (total sleep time/time in bed x 100%). Child (with caregiver assistance) and caregiver complete electronic diaries each morning (~5 mins) during each 1-week assessment and throughout treatment.
Actigraphy - Child | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Primary variables: child sleep onset latency and total sleep time. All other actigraphy variables are secondary. Children wear actigraphs (Fitbit Inspire 3, Google), watch-like device, that monitors light and gross motor activity. Data analyzed using 30s epochs. Validated algorithm estimates SOL, TST, WASO, sleep efficiency and other variables provided by diaries. A combination of diary and actigraphy data estimates bed/waketime variability. Children wear devices 24/7 during each 1-week assessment.
Session Completion | within 1 week post-treatment
  Percentage of treatment sessions completed
Treatment Adherence | within 1 week post-treatment
  Percentage of instructions followed as indicated on treatment adherence logs
Internet Intervention Utility Questionnaire (IIUQ) | within 1 week post-treatment
  16-item measure designed to assess usability, likeability, usefulness, understandability, and convenience of an Internet intervention using a 5-point Likert scale, ranging from 0 (not at all) to 4 (very). Two additional open-ended questions ask about the most and least helpful aspects of the program. Scoring range is 0-64.
Treatment Satisfaction Survey | within 1 week post-treatment
  9-item measure designed to provide feedback on the study, including its structure, assessments, scheduling, working with study staff, and the usability of the intervention platforms using a 10-point Likert scale, ranging from 1 (strongly disagree) to 10 (strongly agree) and open-ended questions
Pediatric Insomnia Severity Index | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Pediatric Insomnia Severity Index is a six-item questionnaire that assesses insomnia symptom severity in children 4-10 years old. Items are rated on a 0-6 point scale based on the child's sleep over the past week. Scoring range is 0-30 with with higher scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
Child Sleep Habits Questionnaire-Abbreviated | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Child Sleep Habits Questionnaire - Abbreviated consists of 22 questions regarding child sleep behaviors on a 1 point scale (0 = never, 7 = always). Higher scores indicating issues with sleep habits.
Pediatric Symptom Checklist-17 | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Pediatric Symptom Checklist-17 is a 17-item questionnaire that measures attention, internalizing, and externalizing problems on a 0-2 scale. Scores range from 0-34 with higher score indicates a greater level of psychosocial impairment.
Behavior Rating Inventory of Executive Function -2nd Edition (BRIEF-2) | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Behavior Rating Inventory of Executive Function -2nd Edition (BRIEF-2) is an 86-item caregiver-report measure of day-to-day executive functioning and impairment. T-scores ranging from 30-90 with higher scores indicating greater executive functioning difficulties
Pediatric Daytime Sleepiness Scale | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Pediatric Daytime Sleepiness Scale is an 8-item questionnaire that measures daytime sleepiness and school-related outcomes on a 5-point scale. Scores range from 0-32 with higher scores indicating greater daytime sleepiness.
Revised Children's Anxiety and Depression Scale-25 | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Revised Children's Anxiety and Depression Scale-25 (caregiver report) is a 25-item scale that measures levels of anxiety and depression on a 4-point scale. Scores range from 0-75 with higher scores indicating more severity in symptoms.
Strengths and Difficulties Questionnaire | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  The Strengths and Difficulties Questionnaire is a 25-item questionnaire that measures five scales (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior) on a 4-point scale. Scores range from 0-40 with higher scores indicating greater difficulties across emotional, behavioral, and peer domains.
Heart rate variability - Child | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  HRV will be assessed using Holter Monitoring during an established stress reactivity protocol. Participants will be seated at rest and undergo Holter Monitoring procedures: 1) 5 min baseline, 2) 30 secs vibrotactile stimuli (Conair WM200X, Stamford, CT) at 80 Hz oscillations applied to left hand, 3) 3 min recovery, 4) 30 secs vibrotactile stimuli applied to right hand, 5) 3 min recovery, 6) cold pressor stimulation to right hand (place hand to bottom of bowl of ice water calibrated to 4° C), 7) 3 min recovery, 8) cold pressor stimulation to left hand. Time and spectral analysis of short-term HRV during baseline, vibration and cold pressor stimuli will be conducted in BioPAC software. Time (reflects beat-to-beat variability-RMSDNN, pNN50) and frequency [reflects underlying HR rhythms-High (0.15-0.4 Hz), low (0.04-0.15 Hz), very low (below 0.04 Hz), LF/HF ratio] domains will be examined.
Peds Quality of Life | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. Caregiver forms will be completed. Scores ranges from 0-100 with higher scores indicating better quality of life.
Heart rate variability - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  HRV will be assessed using Holter Monitoring during an established stress reactivity protocol. Participants will be seated at rest and undergo Holter Monitoring procedures: 1) 5 min baseline, 2) 30 secs vibrotactile stimuli (Conair WM200X, Stamford, CT) at 80 Hz oscillations applied to left hand, 3) 3 min recovery, 4) 30 secs vibrotactile stimuli applied to right hand, 5) 3 min recovery, 6) cold pressor stimulation to right hand (place hand to bottom of bowl of ice water calibrated to 4° C), 7) 3 min recovery, 8) cold pressor stimulation to left hand. Time and spectral analysis of short-term HRV during baseline, vibration and cold pressor stimuli will be conducted in BioPAC software. Time (reflects beat-to-beat variability-RMSDNN, pNN50) and frequency [reflects underlying HR rhythms-High (0.15-0.4 Hz), low (0.04-0.15 Hz), very low (below 0.04 Hz), LF/HF ratio] domains will be examined.
Actigraphy - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Caregiver sleep diary variables include sleep onset latency (lights-out until sleep onset), wake after sleep onset, total sleep time, and sleep efficiency (total sleep time/time in bed x 100%). Caregivers wear actigraphs (Fitbit Inspire 3, Google), a watch-like device that monitors light and gross motor activity. Data analyzed using 30s epochs. Validated algorithm estimates SOL, TST, WASO, sleep efficiency and other variables provided by diaries. A combination of diary and actigraphy data estimates bed/waketime variability. Caregivers wear devices 24/7 during each 1-week assessment.
Electronic Sleep Diaries - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Caregiver sleep diary variables include sleep onset latency (lights-out until sleep onset), wake after sleep onset, total sleep time, and sleep efficiency (total sleep time/time in bed x 100%). Caregiver will complete electronic diaries each morning (~5 mins) during each 1-week assessment and throughout treatment.
State-Trait Anxiety Inventory (STAI-Y1) - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  State-Trait Anxiety Inventory (STAI-Y1) includes 20 self-descriptive statements rated according to how the caregiver generally feels on a 4-point scale [1 (not at all) to 4 (very much so)]. Scores range from 20-80 with higher scores indicate greater levels of anxiety.
Beck Depression Inventory -II - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Beck Depression Inventory (BDI-II) includes 21 items that measures the severity of depressive symptomatology on a 4-point scale (0-absence of symptoms; 3-severe). Scores range from 0-63 with higher scores indicating higher severity of depressive symptoms.
Fatigue Severity Scale - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Fatigue Severity Scale includes 9 items on severity of fatigue and how fatigue interferes with activities on a 7-point scale (1-strongly disagree; 7-strongly agree). Scores range from 9-63 with higher scores indicating severe fatigue symptoms.
Daily Fatigue - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Daily Fatigue rated on electronic diaries (0-none;100-most intense imaginable)
Caregiver Strain Index - Caregiver | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Caregiver Strain Index (CSI) includes 12 items on caregiving impact on well-being. Scoring range 0-26 with higher scores indicate greater caregiver strain

OTHER OUTCOMES:
Pubertal Development Scale (PDS) | baseline, within 1 week post treatment, 1 month follow up, 3 month follow up
  Self-report questionnaire used to assess pubertal status

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided